CLINICAL TRIAL: NCT05114694
Title: Consultant of Shenzhen People's Hospital
Brief Title: Early Arthroscopic Partial Meniscectomy(APM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Hongyu Wang, chief residents, The First People's Hospital of Jingzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APM TIME
Record Dates: First submitted 2021-11-05; First posted 2021-11-10 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early APM (Experimental): Early APM group were patients have knee syndrome within 3 to 6 months
  Interventions: Procedure: early APM
- delayed APM (Placebo Comparator): delayed APM group recruit participants who received delayed APM surgery within 6 to 12 months
  Interventions: Procedure: delayed APM

INTERVENTIONS:
Procedure: early APM — Early APM group were patients have knee syndrome within 3 to 6 months
  Other Names: Early arthroscopic partial meniscectomy
  Arms: early APM
Procedure: delayed APM — delayed APM group recruit participants who received delayed APM surgery within 6 to 12 months
  Other Names: delayed arthroscopic partial meniscectomy
  Arms: delayed APM

SUMMARY:
Arthroscopic partial meniscectomy(APM) surgery outcomes for Metabolic Syndrome(MetS) patients with degenerative meniscus tears(DMTs) was still not clear. The aim of the study was to investigate outcomes of early APM vs delayed APM for MetS patients with degenerate meniscus tears.

DETAILED DESCRIPTION:
Degenerate meniscus tears(DMTs) were the most common knee disease in aged and obese people. The most common treatment for DMTs was arthroscopic partial meniscectomy(APM) surgery. However, the time window for performing APM surgery was unclear, especially in obese patients with Metabolic syndrome(MetS). Abdominal obesity, insulin resistance with or without glucose intolerance, dyslipidemia or elevated blood pressure are included in the principal components of MetS. Whether early APM within 3 to 6 months or delayed APM surgery within 6 to 12 months are benefical to MetS patients with DMTs. The knee function outcomes between early APM and delayed APM for MetS patients with DMTs were assessed and follow up to 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Must be age between 35 and 70 years old;

  * Clinical diagnosis of metabolic syndrome;
  * Clinical diagnosis of degnerate meniscus tears;

Exclusion Criteria:

* Must be able to have no acute knee injury such as car crash or acute sports injury;

  * Must be able to have no knee surgeries history;
  * Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
  * Must be able to have no contraindications to MRI;
  * Must be able to have no severe cardiopulmonary disease;
  * Must be able to have no musculoskeletal or neuromuscular impairments ;
  * Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Knee KOOS score | up to 12 month
  The KOOS was a self-administered outcome questionnaire has been validated in individuals undergoing APM surgery,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
IKDC score | up to 12 month
  The IKDC was a questionnaire that has high reliability and validity for middle to older patients with a meniscal tear,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
waist circumstance | at baseline
  midway between the lowest rib and the iliac crest, using an anthropometric tape
SBP | at baseline
  systolic blood pressure
DBP | at baseline
  diastolic blood pressure
TC | at baseline
  serum total cholesterol (TC)
TG | at baseline
  serum triglycerides (TG)
LDL | at baseline
  serum low-density lipoprotein cholesterol (LDL-C)
HDL | at baseline
  serum high-density lipoprotein cholesterol (HDL-C)
FBG | at baseline
  serum fast blood glucose(FBG)
BMI | at baseline
  BMI, calculated as weight in kilograms divided by height in meters squaredBMI in kg/m^2
K-L grade | at baseline
  Kellgren-Lawrence (K/L) grade

SECONDARY OUTCOMES:
pain score | up to 12 month
  The KOOS subscales for pain,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
symptoms score | up to 12 month
  The KOOS subscales for symptoms,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
activities of daily living score | up to 12 month
  The KOOS subscales for activities of daily living,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
function in sport and recreation score | up to 12 month
  The KOOS subscales for function in sport and recreation,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)
knee related quality of life score | up to 12 month
  The KOOS subscales for knee related quality of life,with 0(extreme knee problem) to 100 points(the best possible score, no knee problems)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning, China